CLINICAL TRIAL: NCT00739258
Title: Surveillance and Medical Help for HIV-infected Intravenous Drug Users in and Out of Prison and Set up the Notional Halfway Home in Union Area of Medical Facility
Brief Title: Surveillance and Medical Help for HIV-infected Intravenous Drug Users in and Out of Prison
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-970077
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections
Keywords: HIV-infected person; Entamoeba; Cryptosporidium; Giardia; ELISA; PCR; IDU; Gonorrhea; Chlamydial trachomatis; Syphilis; Genital warts; Herpes simplex virus
MeSH Terms: conditions — HIV Infections; Giardiasis; Gonorrhea; Syphilis; Condylomata Acuminata; Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIDU: intravenous drug user (IDU) with HIV infected
- IDU: intravenous drug user (IDU) without HIV
- MH: persons receiving methadone maintenance treatment

SUMMARY:
It is difficult to detect the intestinal protozoal infections among the HIV-infected persons or travelers diarrhea by using the traditional microscopy or staining methods. The purpose of this study aimed at finding out the appropriate diagnostic methods and the infection rate of the intestinal protozoa, including the Entamoeba, Cryptosporidium and Giardia among the HIV-infected persons by using the antigen detection method and biological method. The investigators also tried to analyze the associated HIV infection status and sexual transmitted diseases (STD) including Gonorrhea, Chlamydial trachomatis, Syphilis, Genital warts and Herpes simplex virus in this study. The study will collect the blood, urine and stool samples from 200 intravenous drug user (IDU) with HIV-infected in the prisons, 400 intravenous drug user (IDU) without HIV infected and 100 intravenous drug user (IDU) with HIV infected receiving methadone maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV
* Receiving Methadone Maintenance Treatment
* intravenous drug user (IDU)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The samples are obtained from Kaohsiung prison, Kaohsiung women's prison, Pingtung prison and the Kaohsiung Medical University Chung-Ho Memorial Hospital in Kaohsiung, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan